CLINICAL TRIAL: NCT04247386
Title: The Efficacy and Tolerability of Mizone Versus Water in Bowel Preparations: a Randomised Controlled Study
Brief Title: Mizone vs Water for Bowel Preparation.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ningbo No. 1 Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: PEG-1.0
Record Dates: First submitted 2019-12-21; First posted 2020-01-30 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Bowel Preparation
Keywords: bowel preparation quality

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PEG-Mizone prep (Experimental): The evening before the colonoscopy: The patients who are randomized to the " PEG-Mizone prep " arm will drink single dose of 60g Polyethylene Glycol (PEG-4000) with 0.6L Mizone+0.4L water at a rate of 250 ml every 15 min.
  On the day of the colonoscopy: The patients who are randomized to the " PEG-Mizone prep " arm will drink single dose of 120g Polyethylene Glycol (PEG-4000) with 1.2L Mizone+0.8L water 4-6 h before colonoscopy at a rate of 250 ml every 15 min.
  Interventions: Drug: PEG-Mizone
- PEG-ELS prep (Active Comparator): The evening before the colonoscopy: In the PEG-ELS prep group, all the patients drink single dose of 60g Polyethylene Glycol (PEG-4000) with 1L water at a rate of 250 ml every 15 min.
  On the day of the colonoscopy: all the patients drink single dose of 120g Polyethylene Glycol (PEG-4000) with 2L water 4-6 h before colonoscopy at a rate of 250 ml every 15 min.
  Interventions: Drug: PEG-ELS

INTERVENTIONS:
Drug: PEG-Mizone — The evening before the colonoscopy:60gPEG-4000 was mixed with 0.6LMizone and 0.4L water.
  On the day of the colonoscopy:4-6 hours before colonoscopy, 120gPEG-4000 was mixed with 1.2LMizone and 0.8L water.
  Arms: PEG-Mizone prep
Drug: PEG-ELS — The evening before the colonoscopy:60gPEG-4000 was mixed with 1L water. On the day of the colonoscopy:4-6 hours before colonoscopy, 120gPEG-4000 was mixed with 2L water.
  Arms: PEG-ELS prep

SUMMARY:
In order to analyze the effectiveness and patient tolerance of the two bowel preparation regimens, we will compare Polyethylene Glycol Electrolytes Powder (PEG-4000) and Mizone with PEG-ELS. The aim was to demonstrate that polyethylene glycol electrolyte powder (PEG-4000) and Mizone is not inferior in overall quality of intestinal preparation to PEG-ELS in subjects undergoing colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

Patients age between 18-75 years old requiring colonoscopy and willing to participate in this study.

Exclusion Criteria:

1. Patients with constipation;
2. Patients with congestive heart failure;
3. Patients with a history of kidney disease;
4. Patients with a history of poor intestinal preparation;
5. Pregnant / lactating women;
6. Patients without informed consent;
7. Allergic or intolerant to any research drug;
8. Patients with severe gastrointestinal diseases, such as intestinal obstruction or perforation, active ulcerative colitis, toxic colitis and toxic megacolon;
9. Patients with a history of inflammatory bowel disease;
10. Significant electrolyte anomalies, including phosphorus, sodium, potassium, calcium, chloride and magnesium;
11. History of colorectal resection；
12. Patients with diabetes.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2019-12-25 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Quality of Bowel Preparation | 1 Day of colonoscopy
  The OBPS，a scoring system with scores between 0 and 14, where 0 is the best score，divides the colon into 3 segments (right, transverse and rectosigmoid colon); each is scored from 0-4 (0=excellent, If it is necessary to suction liquid stool to adequately see the colonic wall, a score of 2 (fair) is given; if it is necessary to wash and to suction, a score of 3 (poor) is given. The remaining scores fall into place around these anchors. ). A score 0-2 is added to indicate the total amount of luminal fluid.(0=The total amount of fluid in the colon is very small,1=a moderate volume of fluid overall in the colon,2=a large volume of fluid overall in the colon)

SECONDARY OUTCOMES:
Adverse event rate | 3 days
  Including Electrolyte disorders requiring clinical treatment, etc.
patient tolerability of bowel preparation | 1 Day of colonoscopy
  On the day of the patient's colonoscopy, each patient will complete another form regarding their bowel preparation experience with a modified 5-point Likert scale for ease of use (score 5-1: very easy, easy, tolerable, difficult or very difficult).

CONTACTS AND LOCATIONS:
Locations (1):
- Ningbo No. 1 Hospital, Ningbo, Zhejiang, China

REFERENCES:
- [Derived] Zhang Z, Gao H, Yuan X, Liu C, Bao Z, Yu S, Xie H, Wang W, Xie J, Xu L. The efficacy and tolerability of sports drink versus water in bowel preparations: a randomised controlled study. Trials. 2022 Aug 26;23(1):709. doi: 10.1186/s13063-022-06658-2. PMID 36028915